CLINICAL TRIAL: NCT05047484
Title: A Randomized, Double-Blind, Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ACH-0145228 in Healthy Participants
Brief Title: A Study of Multiple Doses of ALXN2050 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ACH228-002
Record Dates: First submitted 2021-09-09; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Healthy
Keywords: Factor D Inhibitor; Complement; ALXN2050; ACH-0145228; Pharmacokinetics; Pharmacodynamics; Safety
MeSH Terms: interventions — rhoA GTP-Binding Protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1: 40 mg ALXN2050/Placebo (Experimental): Participants randomized to receive ALXN2050 or placebo twice daily (BID) on Day 1 through Day 14 in a fasted state.
  Interventions: Drug: ALXN2050; Drug: Placebo
- Cohort 2: 80 mg ALXN2050/Placebo (Experimental): Participants randomized to receive ALXN2050 or placebo BID on Day 1 through Day 14 in a fasted state.
  Interventions: Drug: ALXN2050; Drug: Placebo
- Cohort 3: 120 mg ALXN2050/Placebo (Experimental): Participants randomized to receive ALXN2050 or placebo BID on Day 1 through Day 14 in a fasted state.
  Interventions: Drug: ALXN2050; Drug: Placebo
- Cohort 4: 200 mg ALXN2050/Placebo (Experimental): Participants randomized to receive ALXN2050 or placebo BID on Day 1 through Day 14 in a fasted state.
  Interventions: Drug: ALXN2050; Drug: Placebo
- Cohort 5: 120 mg ALXN2050/Placebo (Experimental): Participants randomized to receive a single dose of ALXN2050 or placebo on Day 1 in a fed state.
  Interventions: Drug: ALXN2050; Drug: Placebo
- Cohort 6: 240 mg ALXN2050/Placebo (Experimental): Participants randomized to receive a single dose of ALXN2050 or placebo on Day 1 in a fasted state.
  Interventions: Drug: ALXN2050; Drug: Placebo

INTERVENTIONS:
Drug: ALXN2050 — Powder-in-capsule (PIC).
  Other Names: ACH-0145228 (formerly); ACH-5228
Drug: Placebo — PIC.

SUMMARY:
This was a Phase 1, placebo-controlled, randomized, double-blind (participant and investigator blind, sponsor open), multiple-ascending dose study conducted in healthy participants to demonstrate the safety and tolerability and to evaluate the pharmacokinetics and pharmacodynamics of ACH-0145228 (ALXN2050).

ELIGIBILITY:
Key Inclusion Criteria:

* Was overtly healthy as determined by medical evaluation including detailed medical history, physical examination, blood pressure and heart rate measurements, 12-lead ECG, and clinical laboratory tests.
* Had a body weight of at least 50 kilograms (kg) and body mass index within the range of 18 to 30 kg/meter squared (inclusive).
* Male participants were eligible to participate if they agreed to abstinence or use of a highly effective method of contraception.
* Female participants must have been of nonchildbearing potential.

Key Exclusion Criteria:

* Had a history or clinically relevant evidence of current cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disorders or conditions capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Had a body temperature greater than or equal to 38°Celsius on Day -1 or Day 1, Hour 0; had a history of febrile illness, or other evidence of infection, within 14 days prior to first study drug administration.
* Had a sensitivity to any of the study interventions, or components thereof, or drug or other allergy that contraindicated participation in the study.
* Donated blood or lost more than 500 milliliters of blood within 3 months prior to first study drug administration, or received a blood transfusion or blood products within 6 months prior to first study drug administration.
* Current enrollment or past participation within the last 30 days before study drug administration in any clinical study involving an investigational study intervention or any other type of medical research
* Had clinically significant laboratory abnormalities.
* Positive urine drug screen at Screening or Day -1; was a current tobacco/nicotine user or smoker; consumed any alcohol within 72 hours before first study drug administration or had a history of regular alcohol consumption within 6 months of screening.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
Number Of Participants Experiencing Serious Adverse Events | Day 1 through Day 42
Number Of Participants Experiencing Grade 3 Or 4 Adverse Events (AEs) | Day 1 through Day 42
Number Of Participants Experiencing AEs Leading To Discontinuation From The Study | Day 1 through Day 42
Number Of Participants Experiencing Grade 3 Or 4 Laboratory Abnormalities | Day 1 through Day 42
Number Of Participants Experiencing Treatment-emergent Vital Signs, Physical Examination Results, And Electrocardiogram (ECG) Abnormalities | Day 1 through Day 42

SECONDARY OUTCOMES:
Maximum Steady-state Plasma Concentration (Cmax,ss) Of Multiple-dose ALXN2050 | Up to 168 hours postdose
Time To Reach Maximum Steady-state Plasma Concentration (Tmax,ss) Of Multiple-dose ALXN2050 | Up to 168 hours postdose
Area Under The Plasma Concentration Versus Time Curve Over The Dosing Interval (AUCtau) Of Multiple-dose ALXN2050 | Up to 168 hours postdose
Maximum Plasma Concentration (Cmax) Of Single-dose ALXN2050 | Up to 72 hours postdose
Time To Reach Maximum Plasma Concentration (Tmax) Of Single-dose ALXN2050 | Up to 72 hours postdose
Area Under The Concentration-time Curve Extrapolated To Infinity (AUC0-inf) For Single-dose ALXN2050 | Up to 72 hours postdose
Alternative Pathway (AP) Activity As Measured By Wieslab Assay | Up to 14 days postdose
Plasma Bb Fragment Of Complement Factor B Concentration Over Time | Up to 14 days postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes